CLINICAL TRIAL: NCT01499160
Title: GCC 0901- A Phase II Study of Letrozole in Combination With Lapatinib Followed by an Addition of Everolimus in Postmenopausal Women With Advanced Endocrine Resistant Breast Cancer
Brief Title: Letrozole and Lapatinib Followed by Everolimus in Women With Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Novartis Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Katherine Tkaczuk, Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040802; GCC 0901; GCC 0901 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2011-12-14; First posted 2011-12-26 (Estimated); Results first posted 2018-03-06 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Breast Neoplasms; Endocrine Breast Diseases; Neoplasm Metastasis
Keywords: endocrine resistant; everolimus; lapatinib; letrozole
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasm Metastasis | interventions — Letrozole; Lapatinib; Everolimus

STUDY DESIGN:
Intervention Model Description: sequential treatment assignment, no masking is done
Masking Description: No masking was done
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HER2-positive or negative (Experimental): Lapatinib 1,500 mg/day + letrozole 2.5 mg/day until progression followed by everolimus 5 mg/day + letrozole 2.5 mg/day + lapatinib 1,250 mg/day.
  Interventions: Drug: letrozole; Drug: lapatinib; Drug: everolimus

INTERVENTIONS:
Drug: letrozole — Drug is are to be taken orally. 2.5 mg once daily
  Other Names: Femara
Drug: lapatinib — Drug is to be taken orally. 1,500 mg once daily in the first part of the study and then 1,250 mg once daily in the second part of the study (after initial progression)
  Other Names: Tykerb
Drug: everolimus — Drug is to be taken orally. 5 mg once daily.
  Other Names: Afinitor

SUMMARY:
About a third of patients with breast cancer are usually treated by hormone pills called tamoxifen and aromatase inhibitors. Aromatase inhibitors are drugs that stop female hormone production. Female hormone or estrogen is an important hormone for the growth of breast cancer cells. Letrozole is one of the aromatase inhibitors that is approved by the FDA and has been used to treat breast cancer since 1997. However, hormone pills usually work for about 6-10 months in most patients. Later on, breast cancer will start to grow again. This condition when hormone pills or endocrine therapy no longer work is called "endocrine resistant" breast cancer. The scientists here at University of Maryland have discovered how these cancer cells can become resistant to hormone pills. In our laboratory tests, the investigators found that lapatinib and everolimus can reverse this resistance and make letrozole work again. However, it is not known if the drugs can reverse the resistance in humans.

The purpose of this study is to find out whether the combination of letrozole, lapatinib, and everolimus is effective in women with breast cancer when hormone pills no longer work.

Lapatinib is an anti-cancer drug that is already approved by the Food and Drug Administration (FDA). It is the standard of care for the treatment of a particular type of breast cancer called human epithelial growth factor receptor 2 (HER2)-positive breast cancer. HER2 is a protein involved in the growth of some cancer cells. This study will also include patients with HER2-negative breast cancer. This means that the cancer cells in these patients do not depend on the HER2 protein. The use of lapatinib in these patients is considered experimental.

Everolimus is also an anti-cancer drug that is approved by the FDA for kidney cancer. Initial studies in mice and later studies in women with breast cancer have shown that everolimus may also slow the growth of breast cancer. The use of everolimus is experimental in this study.

DETAILED DESCRIPTION:
This is a single-institution clinical trial. Patients will be stratified according to the HER2 status:

Group 1: HER2-positive in the tumor tissue Group 2: HER2 negative in the tumor tissue

In the first part of the study, all of the patients will receive the combination of lapatinib 1,500 mg/day and letrozole 2.5 mg/day. We do not expect any significant toxicity from this combination since the previous study of lapatinib and letrozole showed that this combination is safe with no grade 3-4 toxicities observed. Restaging scans (CT scan, MRI, or bone scan) will be obtained after every 12 weeks of treatment. In those patients who progress from any group, everolimus 5 mg/day will be added to letrozole and lapatinib will be reduced to 1,250 mg/day as per the SWOG phase I study of lapatinib and everolimus. The outcome of each group will continue to be assessed separately. We do not expect to see additional serious toxicity from adding everolimus to the combination of lapatinib and letrozole. All of the treatment will be continued until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Female greater than or equal to 18 years.
* Histologically confirmed breast adenocarcinoma with incurable progressing local-regional or metastatic.
* ER and/or PR positivity of primary and/or secondary tumor.
* Patients must have measurable or evaluable disease.
* Evidence of disease progression or relapse while on or less than 6 months off aromatase inhibitors or tamoxifen either in adjuvant or first line metastatic setting.
* Postmenopausal
* Patients may have received up to one prior chemotherapy regimen for stage IV breast cancer. Prior chemotherapy in the adjuvant and/or neoadjuvant setting is permitted. Chemotherapy must be finished at least 2 weeks prior to enrollment.
* ECOG performance status <2
* Fasting cholesterol ≤300 mg/dL OR ≤7.75 mmol/LAND fasting triglycerides ≤ 2.5 x ULN despite appropriate treatment.
* Patients must have adequate organ function as defined by the protocol.
* Stratification 1:

  * HER2 positive in the primary or secondary tumor tissue
  * Prior trastuzumab therapy is allowed but NOT required. However, trastuzumab should be discontinued at least 3 weeks prior to enrollment.
* Stratification 2:

  * HER2 negative in the primary or secondary tumor tissue

Exclusion Criteria:

* Patients receiving any other investigational agents.
* Prior exposure to lapatinib, everolimus, or other mTOR inhibitors.
* History of allergic reactions or hypersensitivity to compounds similar to everolimus, lapatinib, or letrozole.
* Patients who have any severe and/or uncontrolled medical conditions that could affect their participation such as:

  * Left ventricular ejection fraction (LVEF) < 50%
  * Unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
  * Severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is ≤ 88% at rest on room air.
  * Uncontrolled diabetes
  * Active or uncontrolled severe infection
* Patients with QTc interval > 0.47 seconds.
* Significant chronic or acute gastrointestinal disorder with diarrhea as a major symptom.
* Prior exposure to more than 360 mg/m2 doxorubicin, more than 120 mg/m2mitoxantrone, or more than 90 mg/m2idarubicin, or elevated baseline cardiac troponin I.
* Patients with active CNS metastasis and/or carcinomatous meningtitis. However, patients with CNS metastasis who have completed a therapy and are clinically stable for 3 weeks as defined as: (1) no evidence of new or enlarging CNS metastasis and (2) off steroids and/or anticonvulsants.
* Patient is known to be HIV, Hepatitis B, or Hepatitis C-positive (these tests are not required).
* Patients with current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease).
* Patients with INR ≥ 2 or PTT ≥ 2 x upper normal limit.
* Previous or current systemic malignancy other than breast cancer within the past 3 years other than carcinoma in situ of the cervix or basal/squamous carcinoma of the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tkaczuk, MD, Principal Investigator — University of Maryland Marlene & Stewart Greenebaum Cancer Center
Locations (1):
- University of Maryland Marlene & Stewart Greenebaum Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University Medical Centers and Hospital Based Oncology Programs recruited participants from July 2012 to December 2014.
Pre-assignment Details: All 7 patients (2 pts were HER2+ and 5 pts were HER2-) started the combination of lapatinib 1,500 mg/day and letrozole 2.5 mg/day.
Groups:
- Letrozole in Combination With Lapatinib Followed by Everolimus: Group 1: HER2-positive in the tumor tissue Group 2: HER2 negative in the tumor tissue
  In the first part of the study, all of the patients will receive the combination of lapatinib 1,500 mg/day and letrozole 2.5 mg/day. Restaging scans (CT scan, MRI, or bone scan) will be obtained after every 12 weeks of treatment. In those patients who progress from any group, everolimus 5 mg/day will be added to letrozole and lapatinib will be reduced to 1,250 mg/day as per the SWOG phase I study of lapatinib and everolimus.
  letrozole: Drug is are to be taken orally. 2.5 mg once daily
  lapatinib: Drug is to be taken orally. 1,500 mg once daily in the first part of the study and then 1,250 mg once daily in the second part of the study (after initial progression)
  everolimus: Drug is to be taken orally. 5 mg once daily.
Period: Overall Study
Arm/Group | Letrozole in Combination With Lapatinib Followed by Everolimus
Started | 7
Completed (number of who completed all study treatments) | 5 (1 pt-withdrew consent 1pt-had cardiac toxicity)
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Letrozole in Combination With Lapatinib Followed by Everolimus
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] — age is a continuous variable and is collected from patient's charts
  years | 60 [50 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate of Patients Treated With the Combination of Letrozole and Lapatinib and Then After Progression, Treated With Everolimus, Letrozole and Lapatinib.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
  Clinical benefit rate is defined as complete response+partial response+ stable disease. All participants will be treated with the combination of letrozole and lapatinib. Once the participant progresses on this regimen, the participant will be treated with everolimus, letrozole and lapatinib until they progress.
Time Frame: From date of study entry until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Population: 1 patient withdrew during cycle 1
Measure: Count of Participants; unit: Participants
Groups:
- Letrozole in Combination With Lapatinib Followed by Everolimus: Group 1: HER2-positive in the tumor tissue-2 subjects Group 2: HER2 negative in the tumor tissue-5 subjects
  In the first part of the study, all of the patients will receive the combination of lapatinib 1,500 mg/day and letrozole 2.5 mg/day. Restaging scans (CT scan, MRI, or bone scan) will be obtained after every 12 weeks of treatment. In those patients who progress from any group, everolimus 5 mg/day will be added to letrozole and lapatinib will be reduced to 1,250 mg/day as per the SWOG phase I study of lapatinib and everolimus.
  letrozole: Drug is are to be taken orally. 2.5 mg once daily
  lapatinib: Drug is to be taken orally. 1,500 mg once daily in the first part of the study and then 1,250 mg once daily in the second part of the study (after initial progression)
  everolimus: Drug is to be taken orally. 5 mg once daily.
Arm/Group | Letrozole in Combination With Lapatinib Followed by Everolimus
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: PROGRESSION FREE SURVIVAL TUMOR ASSESSMENT
Description: Patients treated with the combination of Letrozole and Lapatinib will provide tumor biopsy sample
Time Frame: From date of study entry until 4 weeks after removal from study or until death (whichever occurs first) up to 24 months.
Population: data analysis was not conducted due to low sample (low accrual) and study closure
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole in Combination With Lapatinib Followed by Everolimus
Number analyzed (Participants) | 6
Participants | 6
Statistical Analysis 1: Comparison: Letrozole in Combination With Lapatinib Followed by Everolimus; Not done due to low accrual; Test type: Other — Not done due to low accrual; Not done due to low accrual — Not done due to low accrual; Not done due to low accrual; Not done due to low accrual

ADVERSE EVENTS:
Time Frame: Adverse events including serious adverse events (SAEs) were collected from the start of study until 30 days after completion of last study drug dose on all study patients (7), but only 4 severe adverse events were noted as reported previously.
Arm/Group | Letrozole in Combination With Lapatinib Followed by Everolimus
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole in Combination With Lapatinib Followed by Everolimus (N=7)
Decreased LVEF (Blood and lymphatic system disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
rectal pain (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole in Combination With Lapatinib Followed by Everolimus (N=7)
abdominal pain (Gastrointestinal disorders) | 2 (2)
accidental everolimus overdose (Injury, poisoning and procedural complications) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 2 (2)
arthralgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
dehydration (General disorders) | 1 (1)
diaphoresis (General disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 5 (11)
dizziness (General disorders) | 2 (2)
elevated ALT & AST (Endocrine disorders) | 5 (9)
epigastric pain (Gastrointestinal disorders) | 1 (1)
epistaxis (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (8)
Fracture fibula (Musculoskeletal and connective tissue disorders) | 1 (1)
hair loss (General disorders) | 2 (2)
hip pain (Musculoskeletal and connective tissue disorders) | 2 (2)
hypertriglyceridemia (General disorders) | 2 (2)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leucopenia (Blood and lymphatic system disorders) | 1 (2)
lymphedema (Blood and lymphatic system disorders) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
mouth ulcers (General disorders) | 1 (1)
mucositis (General disorders) | 3 (6)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (6)
numbness in toes (General disorders) | 1 (1)
Otitis Externa (Ear and labyrinth disorders) | 1 (1)
pain (General disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 5 (10)
right back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
right eyelid swelling (Eye disorders) | 1 (1)
right foot pain (General disorders) | 1 (1)
right hip pain (General disorders) | 1 (1)
right shoulder pain (General disorders) | 1 (1)
right toe cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
righted sided pain (General disorders) | 1 (1)
stomatitis (General disorders) | 1 (1)
URI (Respiratory, thoracic and mediastinal disorders) | 2 (2)
UTI (Renal and urinary disorders) | 1 (1)
vomiting (General disorders) | 1 (1)
weight gain (General disorders) | 1 (1)
weight loss (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes